CLINICAL TRIAL: NCT03103802
Title: Evaluation of the Accuracy of Digital Models Obtained Using Intraoral and Extraoral Scanners Versus Gold Standard Plaster Model (Diagnostic Accuracy Study)
Brief Title: Evaluation of the Accuracy of Digital Models Obtained Using Intraoral and Extraoral Scanners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moahmed Amr Labib, Intern Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CEBD-CU-2017-03-24
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Orthodontics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intra-oral scanning (Experimental)
  Interventions: Device: intra-oral digital scanner and extra-oral digital scanner
- extra-oral scanning of the plaster model obtained via alginate (Experimental)
  Interventions: Device: intra-oral digital scanner and extra-oral digital scanner
- extra-oral scanning of plaster model obtained via rubber base (Experimental)
  Interventions: Device: intra-oral digital scanner and extra-oral digital scanner
- extra-oral scanning of the rubber base impression (Experimental)
  Interventions: Device: intra-oral digital scanner and extra-oral digital scanner
- extra-oral scanning of the alginate impression (Experimental)
  Interventions: Device: intra-oral digital scanner and extra-oral digital scanner

INTERVENTIONS:
Device: intra-oral digital scanner and extra-oral digital scanner — intra-oral and extra-oral digital scanners used to obtain digital models

SUMMARY:
This study is to compare the diagnostic accuracy of digital models obtained via 10 digitization techniques to the reference standard of orthodontic plaster model through dental measurements

ELIGIBILITY:
Inclusion Criteria:

* adult patients seeking orthodontic treatment permanent dentition

Exclusion Criteria:

* deciduous or mixed dentition cleft lip and palate patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-04-30 (Estimated); Primary Completion 2017-10-30 (Estimated); Study Completion 2018-02-27 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 6 months
  evaluation of the accuracy of digital models obtained using scanners

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Hazem, PHD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry- Cairo University, Cairo Governorate, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes